CLINICAL TRIAL: NCT02290405
Title: Impact of Hyperarousal on Simple and Complex Cognitive Task Performance Among Insomnia Sufferers
Status: Completed | Type: Observational
Sponsor: Jack Edinger, PhD (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Jack Edinger, PhD, Professor, Department of Medicine, National Jewish Health
Organization: National Jewish Health (Other)
Other Study IDs: 2786
Record Dates: First submitted 2014-11-04; First posted 2014-11-14 (Estimated); Results first posted 2021-03-30 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2018-05

CONDITIONS: Insomnia; Primary Insomnia; Chronic Insomnia
Keywords: insomnia; primary insomnia; chronic insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Primary Insomnia (PI): PI sufferers enrolled will meet Research Diagnostic Criteria for insomnia disorder, score > 14 on the Insomnia Severity Index, report insomnia for > 3 months, have sleep difficulties > 3 nights per week, score < 3 on the Epworth Sleepiness Scale (ESS), score > 40 on the Hyperarousal Scale10 and report an inability to nap in the daytime.
  Interventions: Behavioral: Multiple Sleep Latency Test (MSLT)
- Normal Sleepers (NS): The normal sleepers enrolled will report general satisfaction with sleep and no sleep/wake complaints, score < 10 on the ESS, score < 35 on the Hyperarousal Scale10, and deny a practice of routine daytime napping.
  Interventions: Behavioral: Multiple Sleep Latency Test (MSLT)

INTERVENTIONS:
Behavioral: Multiple Sleep Latency Test (MSLT) — The daytime protocol will include a 4-trial Multiple Sleep Latency Test (MSLT) along with 4-trials of a computer -administered battery of reaction time tasks. The assessment protocol will start two to three hours after participants' respective morning rising times and will begin with a battery of the neuro-cognitive testing followed by an MSLT nap. Per standard MSLT procedures, the daytime testing will be scheduled so the four performance testing and sleepiness assessment trials occur two hours apart. All daytime testing will be conducted under the supervision of trained laboratory technologists.

SUMMARY:
The purpose of this study is to learn more about people with insomnia disorder and cognitive impairment. Cognitive impairment is difficulty with mental abilities such as thinking, knowing and remembering.

DETAILED DESCRIPTION:
Primary insomnia (PI) sufferers typically complain of such daytime impairments as reduced attention, concentration, memory and global mental acuity. Moreover, epidemiological studies have shown PI contributes to reduced productivity, work and traffic accidents, and serious falls among the elderly. Despite such findings, laboratory-based efforts to corroborate the cognitive complaints of PI sufferers have produced mixed results. Indeed, many studies comparing PI sufferers with non-complaining normal sleepers across a range of neuropsychological tests have failed to show any relative deficits among the PI group. Such findings, in turn, has led to the impression that PI patients cognitive complaints may be over-stated and result from their attentional bias toward minor cognitive errors, dysfunctional beliefs about the impact of insomnia on functioning or excessive self focus rather than to any measurable daytime impairment.

However, many previous such studies were underpowered due to small sample sizes and employed neuropsychological tests designed for detecting impairment resulting from brain disease/damage rather than the more subtle albeit significant impairments of which PI patients complain. In recent research, we and others have shown that PI sufferers do, indeed, show greater deficits (slower and more variable reaction times) particularly on complex switching attention tasks. Moreover, there is some preliminary evidence that the subgroup of PI sufferers with elevated levels of physiological hyperarousal are most prone to suffer from neuro-cognitive performance deficits than are matched groups of PI sufferers who are not physiologically hyperaroused and normally alert individuals without insomnia. For example, Fernandez-Mendoza recently showed that PI sufferers with a hyperarousal pattern suggested by their objective short sleep duration on serial polysomnograms (PSG) performed more poorly on a complex switching attention task than did both normal sleepers and PI sufferers with normal objective sleep durations.

In our efforts to follow up on this latter work, we recently examined the error rates of alert and sleepy PI sufferers and normal sleepers across a series of simple and complex reaction time tasks. We employed age and gender matched samples of PI (N=89) sufferers and normal sleepers-NS (N=95). Participants underwent three nights of PSG followed by daytime testing with a four-trial Multiple Sleep Latency Test-MSLT. The PI and NS groups were each subdivided into "alert" (e.g., MSLT mean onset latency > 8 minutes) and "sleepy" (e.g., MSLT mean onset latency < 8 minutes) subgroups to allow for testing the main and interaction effects of participant type and level of alertness. "Alert" participants had longer MSLT latencies than "sleepy" participants (12.7 vs. 5.4 minutes). PI sufferers had fewer correct responses on performance testing than did NS. However, as shown by the adjacent, figure we found a significant group x alertness interaction (p = .0013) with greater error rates occurring among alert (hyperaroused) PI sufferers (Mean=4.5±3.6 errors per trial) than among alert NS (Mean=2.6±1.9 errors per trial). This was particularly true for the more complex switching attention task.

Our work along with that of Fernandez-Mendoza serve to confirm that PI sufferers have measureable objective neuro-cognitive deficits and provide some preliminary suggestion for the types of testing approaches that should be used to detect them. The identification of tests sensitive to PI sufferers' cognitive deficits are particularly relevant for testing the effects of current and future insomnia therapies on patients' objective daytime functioning. Measures of daytime dysfunction can and should serve as endpoints for assessing benefits and detriments of insomnia therapies. In addition, our recent work suggests that subgroups of PI sufferers may differ in their daytime deficits, with those showing physiological hyperarousal being most prone to make errors. This finding suggests that different types or doses of treatment may be needed to reverse the daytime impairments of the hyperaroused and non-aroused PI patients. However, our line of research would benefit by replication and extension findings to (1) further confirm the detrimental effects of physiological hyperarousal on PI sufferer's neuro-cognitive functioning; and (2) identify a broader range of tests that can be used for assessing diurnal cognitive impairments in both physiologically hyperaroused and lesser aroused PI groups. The current project will address these aims.

ELIGIBILITY:
Inclusion Criteria:

* 21 to 80 years of age
* Insomnia sufferers enrolled, will meet Research Diagnostic Criteria for insomnia disorder
* score > 14 on the Insomnia Severity Index
* report insomnia for > 3 months
* have sleep difficulties > 3 nights per week
* score < 3 on the Epworth Sleepiness Scale (ESS)
* score > 40 on the Hyperarousal Scale and report an inability to nap in the daytime
* The normal sleepers enrolled will report general satisfaction with sleep and no sleep/wake complaints, score < 10 on the ESS, score < 35 on the Hyperarousal Scale, and deny a practice of routine daytime napping

Exclusion Criteria:

* sleep-disruptive medical condition (e.g., rheumatoid arthritis)
* current major psychiatric (Axis I) condition on the basis of a Structured Clinical Interview for Psychiatric Disorders (SCID)
* sedative hypnotic dependence and unwillingness/inability to abstain from these medications while in the study
* use of anxiolytics, antidepressants, or any other psychotropic medication
* an apnea/hypopnea index (AHI) > 5 or a periodic limb movement-related arousal index > 5 during on screening PSG that includes a full sleep montage to allow for detection/diagnosis of sleep-disordered breathing and Periodic Limb Movement Disorder (PLMD).
* female participants who have tested positive on urine pregnancy tests or planing on becoming pregnant during the study
* Additionally, self-described NS who meet criteria for any sleep disorder and those insomnia sufferers who meet criteria for a comorbid sleep disorder in addition to insomnia disorder will also be excluded

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will use a matched-groups cross-sectional experimental design. Age and gender matched groups of hyperaroused PI sufferers and non-complaining normal sleepers (NS) will be recruited and enrolled. A comprehensive screening process that includes structured sleep and psychiatric interviews, screening questionnaires, medical exam, and diagnostic PSG will be used to determine eligible subjects.
Sampling Method: Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jack Edinger, PhD, Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health, Denver, Colorado, United States

REFERENCES:
- [Derived] Edinger JD, Bathgate CJ, Tsai S, Khassawneh B. Impact of daytime sleepiness and insomnia on simple and complex cognitive task performances. Sleep Med. 2021 Nov;87:46-55. doi: 10.1016/j.sleep.2021.08.004. Epub 2021 Aug 12. PMID 34509774

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Primary Insomnia (PI) | Normal Sleepers (NS)
Started | 36 | 53
Completed | 35 | 53
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Primary Insomnia (PI) sufferers enrolled met Research Diagnostic Criteria for insomnia disorder and normal sleepers enrolled reported general satisfaction with sleep and no sleep/wake complaints.
Groups:
- Total: Total of all reporting groups
Arm/Group | Primary Insomnia (PI) | Normal Sleepers (NS) | Total
Number analyzed (Participants) | 36 | 53 | 89
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 52 | 85
  >=65 years | 3 | 1 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.6 (14.1) | 31.5 (10.5) | 35.1 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 37 | 63
  Male | 10 | 16 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 7
  Not Hispanic or Latino | 34 | 48 | 82
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 32 | 46 | 78
  More than one race | 1 | 4 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 36 | 53 | 89

OUTCOME MEASURES:

1. Primary Outcome: Number of Incorrect Trials During the Computer-administered Attention-Switching Task Test.Attention-Switching Task Latency Error Rate
Description: Number of incorrect trials during the computer-administered Attention-Switching Task test, aka Attention-Switching Task test.Attention-Switching Task Latency Error Rate
Time Frame: All study activities for each participant were conducted during a one-day period
Measure: Mean (97.5% Confidence Interval); unit: trials
Arm/Group | Primary Insomnia (PI) | Normal Sleepers (NS)
Number analyzed (Participants) | 35 | 53
trials | 5.11 [4.26 to 5.96] | 3.1 [2.39 to 3.817]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from study start to study completion (up to two days).
Description: No study-related adverse events occurred.
Arm/Group | Primary Insomnia (PI) | Normal Sleepers (NS)
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/53
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/53
Other Adverse Events (participants affected / at risk) | 0/36 | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-05-18): https://cdn.clinicaltrials.gov/large-docs/05/NCT02290405/Prot_SAP_000.pdf